CLINICAL TRIAL: NCT05645783
Title: Liquid Biopsy for Early DiagNosis of Squamous Cell Carcinoma of the HeAd and NeCk rEgion (ENHANCE Study)
Brief Title: Liquid Biopsy for Early DiagNosis of Squamous Cell Carcinoma of the HeAd and NeCk rEgion
Acronym: ENHANCE
Status: Recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5610
Record Dates: First submitted 2022-10-28; First posted 2022-12-12 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A 20ml blood sample (2x 10ml blood collection tube, Streck or other appropriate) for plasma extraction and collection of buffy coat or PBMCs will be taken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The 5-year survival for Head and Neck squamous cell carcinoma (HNSCC) across all TNM stage groups is approximately 50%. Patients who are present with stage I & II disease have significantly better survival. When a patient presents to their general practitioner (GP) with symptoms suggestive of HNSCC, they may be referred for urgent specialist input through the suspected cancer referral (SCR) pathway, which include dedicated neck lump clinics. HNSCC is known to shed fragments of DNA, called circulating tumor DNA (ctDNA) into the bloodstream. The investigators have developed novel ultra-sensitive (>90% sensitivity) next generation sequencing (NGS) assay for circulating HPV DNA in patients with non-metastatic locally advanced head and neck cancer. The use of ultra-sensitive NGS assay for detection of ctDNA using a simple blood test (liquid biopsy) holds a great promise for cancer screening and early diagnosis and can lead to better survival results and less disease burden. With a quicker turnaround (1-2 weeks), the liquid biopsy can help expedite the patient journey through the cancer pathways reducing the incidence of cancer target breaches. In order to design studies to test this hypothesis the investigators require preliminary data quantifying sensitivity and specificity of the assay in this setting.

DETAILED DESCRIPTION:
The 5-year survival for Head and Neck squamous cell carcinoma (HNSCC) across all TNM stage groups is approximately 50%. Patients who are present with stage I & II disease have significantly better survival. When a patient presents to their general practitioner (GP) with symptoms suggestive of HNSCC, they may be referred for urgent specialist input through the suspected cancer referral (SCR) pathway, which include dedicated neck lump clinics. Majority of the patients diagnosed via the SCR pathway present with Stage III &IV disease, which has a direct impact on outcomes.

HNSCC is classified as an uncommon cancer and as such diagnosis and treatment is undertaken in specialist tertiary referral centres. The care of patients initially diagnosed with HNSCC in smaller secondary care hospitals is transferred to these specialist tertiary referral centres via the Inter Trust Transfer (ITT). ITT can introduce delays in treatment pathways resulting in a failure to achieve cancer treatment targets. Southwest London HNSCC diagnostic pathway review which was undertaken in February 2021 demonstrated that 40% of ITTs received were greater than 38 days after referral and that 68% of the 62 day target breaches were in patients with ITT.

HNSCC is known to shed fragments of DNA, called circulating tumor DNA (ctDNA) into the bloodstream. The investigators have developed novel ultra-sensitive (>90% sensitivity) next generation sequencing (NGS) assay for circulating HPV DNA in patients with non-metastatic locally advanced head and neck cancer. The investigator's current work involves ctDNA detection to cover the spectrum of genetic alterations in HNC using a single sequencing workflow to detect copy number aberrations (CNAs), HPV DNA (to cover 99.9% of HNC related HPV) and somatic mutations.

The use of ultra-sensitive NGS assay for detection of ctDNA using a simple blood test (liquid biopsy) holds a great promise for cancer screening and early diagnosis and can lead to better survival results and less disease burden. This has been proven in proof of principle studies in nasopharyngeal cancer (Chan N Engl J Med 2017; 377:513-522). Furthermore, this test can be administered in smaller secondary care hospitals in parallel to the ITT. With a quicker turnaround (1-2 weeks), the liquid biopsy can help expedite the patient journey through the cancer pathways reducing the incidence of cancer target breaches. In order to design studies to test this hypothesis the investigators require preliminary data quantifying sensitivity and specificity of the assay in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for an Ultrasound guided fine needle aspiration (USFNA) in the neck lump clinic

Exclusion Criteria:

* Patient found to have a lump in the thyroid gland at the time of USFNA
* Unable to give informed consent for biological sample collection
* Unable to safely participate in clinic sample collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the neck lump clinics via the SCR pathway, who are classified as high risk and referred for an USFNA.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Measure the sensitivity of the NGS assay for detection of ctDNA in patients with early HNSCC | 1 year

SECONDARY OUTCOMES:
Measure the specificity of the NGS assay for detection of ctDNA at baseline in patients with early HNSCC | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Kingston Hospital Foundation Trust, Kingston upon Thames
  - Northwick Park Hospital, London

REFERENCES:
- [Background] https://www.cancerresearchuk.org/health-professional/cancer-statistics/statistics-by-cancer-type/head-and-neck-cancers.
- [Background] Lee JY, Garcia-Murillas I, Cutts RJ, De Castro DG, Grove L, Hurley T, Wang F, Nutting C, Newbold K, Harrington K, Turner N, Bhide S. Predicting response to radical (chemo)radiotherapy with circulating HPV DNA in locally advanced head and neck squamous carcinoma. Br J Cancer. 2017 Sep 5;117(6):876-883. doi: 10.1038/bjc.2017.258. Epub 2017 Aug 15. PMID 28809864
- [Background] Lam WKJ, Jiang P, Chan KCA, Cheng SH, Zhang H, Peng W, Tse OYO, Tong YK, Gai W, Zee BCY, Ma BBY, Hui EP, Chan ATC, Woo JKS, Chiu RWK, Lo YMD. Sequencing-based counting and size profiling of plasma Epstein-Barr virus DNA enhance population screening of nasopharyngeal carcinoma. Proc Natl Acad Sci U S A. 2018 May 29;115(22):E5115-E5124. doi: 10.1073/pnas.1804184115. Epub 2018 May 14. PMID 29760067

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/83/NCT05645783/Prot_SAP_000.pdf